CLINICAL TRIAL: NCT04858776
Title: Perivenous Dexamethasone Therapy: Examining Reduction of Inflammation After Thrombus Removal to Yield Benefit in Subacute and Chronic Iliofemoral DVT (DEXTERITY-SCI)
Brief Title: Perivenous Dexamethasone Therapy: Examining Reduction of Inflammation After Thrombus Removal to Yield Benefit in Subacute and Chronic Iliofemoral DVT
Acronym: DEXTERITY-SCI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mercator MedSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIP0218
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Iliofemoral; Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment (Experimental)
  Interventions: Combination Product: Perivascular dexamethasone
- Control (Sham Comparator)
  Interventions: Combination Product: Perivascular sham

INTERVENTIONS:
Combination Product: Perivascular dexamethasone — Dexamethasone delivery around target vein segment(s)
  Arms: Treatment
Combination Product: Perivascular sham — Saline delivery around target vein segment(s)
  Arms: Control

SUMMARY:
This is a study of a medical procedure that utilizes a commercially available catheter (the Bullfrog® Micro-Infusion Device) to locally deliver a commercially available anti-inflammatory drug (dexamethasone sodium phosphate injection) around the deep veins after DVT recanalization, where DVT symptoms were present for at least 14 days and no more than 60 days prior to recanalization. The goal of the study is to see if local anti-inflammation helps prevent re-thrombosis of the blood vessel and improvement in symptoms for up to 24 months after the initial DVT recanalization procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form prior to receiving any non-standard of care, protocol-specific procedures.
2. Stated willingness to comply with all study procedures including completion of questionnaires and follow-up visits and availability for the duration of the study.
3. Male or female, aged 18 to 89 years.
4. For females of reproductive potential: negative pregnancy test ≤7 days before the procedure, use of highly effective contraception for at least 1 month prior to screening, and agreement to use such a method during study participation.
5. Negative COVID-19 test result within 5 days prior to procedure or evidence of COVID-19 vaccine or booster within past 12 months.
6. Onset of DVT symptoms 14 to 60 days prior to intervention in the study limb with need for stenting of the iliofemoral segment.
7. Ability to take oral medication and be willing to adhere to the prescribed anti-coagulant regimen.
8. Prescription for at least 14 days low molecular weight heparin followed by therapeutic anticoagulant of investigator's choice for 12-month minimum as part of post-interventional medication regimen.
9. Minimum of 30 days of prescribed antiplatelet agent (aspirin or P2Y12 inhibitor).
10. Hemodynamically significant DVT (>50% area obstruction) spanning at least (a) the iliofemoral and common femoral veins or (b) the common femoral vein with extension into the femoral vein and/or profunda vein. Extent of thrombus in the popliteal and calf veins is allowed.
11. Successful recanalization of the target vein with at least one patent inflow vein (femoral or profunda).

Exclusion Criteria:

1. Current enrollment in another non-registry clinical study of systemic drug therapy or another device study that has not completed its primary endpoint, including prior enrollment in this study. Concurrent enrollment in registry studies of approved devices or drugs are acceptable.
2. Lack of capability of understanding the nature, significance and implications of the clinical trial.
3. Body Mass Index > 40 kg/m2.
4. Non-ambulatory status prior to DVT occurrence.
5. In the target vein segment: previously treated symptomatic DVT within the previous 12 months.
6. In the contralateral (non-study) leg: symptomatic DVT that, in the opinion of the operating physician, will require surgery in the following 30 days.
7. Limb-threatening circulatory compromise with ankle-brachial index <0.4, absolute ankle pressure <50 mmHg or absolute toe pressure <30 mmHg.
8. Pulmonary embolism (PE) defined as either massive (Systolic blood pressure < 90 mmHg and/or patient on IV vasoactive medication to support blood pressure), or intermediate high-risk PE, as defined by the European Society Guideline on management of PE. Low-risk PE and/or intermediate low-risk PE can be enrolled.
9. Inability to tolerate contemporary venous intervention procedure due to severe dyspnea or acute systemic illness.
10. Allergy, hypersensitivity, or thrombocytopenia from heparin, Recombinant tissue plasminogen activator (rtPA), dexamethasone sodium phosphate or iodinated contrast, except for mild-moderate contrast allergies for which steroid pre-medication can be used.
11. History of, or active heparin-induced thrombocytopenia (HIT).
12. Haemoglobin < 9.0 mg/dl, INR > 1.6 before starting anticoagulation, or platelets < 100,000/ml. Moderate renal impairment in diabetic patients (estimated glomerular filtration rate < 60 ml/min) or severe renal impairment in non-diabetic patients (estimated glomerular filtration rate < 30 ml/min).
13. Active bleeding, recent (< 3 mo) GI bleeding, severe liver dysfunction, bleeding diathesis.
14. Recent (< 3 mo) internal eye surgery or haemorrhagic retinopathy; recent (< 10 days) major surgery, cataract surgery, trauma, cardiopulmonary resuscitation, obstetrical delivery, or other invasive procedure.
15. History of hemorrhagic stroke or intracranial/intraspinal bleed, tumor, vascular malformation, aneurysm.
16. Active cancer with a life expectancy of <2 years.
17. Severe hypertension on repeated readings (systolic blood pressure > 180 mmHg or diastolic blood pressure > 105 mmHg). This can be treated, and blood pressure must be stable before venous access is obtained (systolic blood pressure <140 mmHg).
18. Pregnant or breastfeeding.
19. Life expectancy < 2 years.
20. Thrombus of the inferior vena cava (IVC) extending at least one centimeter above the common iliac confluence.
21. Inability to obtain venous access.
22. Inability to recanalize the target vein segment(s).
23. History of ipsilateral venous stent.
24. DVT length to be targeted for perivascular drug therapy exceeds 50 cm.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinically relevant primary patency | 6 months
  Freedom from loss of patency with associated symptoms
Freedom from major adverse event (MAE) | 30 days
  Freedom from composite of all-cause death, clinically significant pulmonary embolism, major bleeding, target vessel thrombosis, infection of treatment or insertion site, or AV fistula of treatment site

CONTACTS AND LOCATIONS:
Locations (15):
- United States (13):
  - Vascular Care Connecticut, Darien, Connecticut
  - University of South Florida, Tampa, Florida
  - Northwestern University Hospital, Chicago, Illinois
  - CIS Clinical Research, Houma, Louisiana
  - Medstar Health Research Institute, Hyattsville, Maryland
  - Stony Brook University Hospital, Stony Brook, New York
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - OhioHealth Research Institute, Columbus, Ohio
  - St John Health System, Bartlesville, Oklahoma
  - CardioVoyage, Denison, Texas
  - University of Texas, Houston, Houston, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Lake Washington Vascular, Bellevue, Washington
- Galway University Hospital, Galway, Ireland
- Guy's and St. Thomas Hospital, London, United Kingdom